CLINICAL TRIAL: NCT07316166
Title: Comparison of Suprainguinal Fascia Iliac Block With and Without Dexmedetomidine as an Adjunct to Ropivacaine for Postoperative Analgesia Following Hip Surgery: a Randomized, Double-blinded Study.
Brief Title: Suprainguinal Fascia Iliaca Block With vs Without Dexmedetomidine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Vendhan Ramanujam, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2264738
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management
Keywords: Hip Surgery; Nerve block
MeSH Terms: interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ropivacaine (Active Comparator): 30 ml of 0.25% ropivacaine; No dexmedetomidine
  Interventions: Drug: Ropivacaine
- Ropivacaine plus Dexmedetomidine (Experimental): 30 ml of 0.25% ropivacaine; 1 mcg/kg of dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Participants in the experimental arm receive a preoperative suprainguinal fascia iliaca block consisting of 30 mL of 0.25% ropivacaine combined with perineural dexmedetomidine at a dose of 1 mcg/kg.
  Arms: Ropivacaine plus Dexmedetomidine
Drug: Ropivacaine — In the experimental arm, ropivacaine (30 mL of 0.25%) is administered with dexmedetomidine.
  In the active comparator arm, ropivacaine (30 mL of 0.25%) is administered alone without any dexmedetomidine medication.

SUMMARY:
The investigators are evaluating postoperative outcomes in patients undergoing hip replacement surgery performed with either spinal or general anesthesia, who also receive a suprainguinal fascia iliaca block using either perineural ropivacaine alone or ropivacaine combined with dexmedetomidine.

DETAILED DESCRIPTION:
Patients undergoing hip replacement surgery often receive a single-shot suprainguinal fascia iliaca block as a part of the primary anesthetic and multimodal postoperative analgesic strategy. However, the analgesic effect of a single-shot block typically diminishes after several hours and may be inconsistent beyond 24 hours. Adding dexmedetomidine, an alpha-2 agonist, to the local anesthetic has been shown to prolong block duration and reduce postoperative opioid requirements. Investigating its use in suprainguinal fascia iliaca blocks for total hip arthroplasty may clarify its clinical effectiveness. The investigators hypothesize that patients receiving ropivacaine with dexmedetomidine will have a significantly longer time to first analgesic request compared to those receiving ropivacaine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total hip arthroplasty
* 18-80 years old
* ASA 1-3 classifications

Exclusion Criteria:

* ASA classification of 4 or greater
* Infection at the site of nerve blockade
* Coagulopathy
* Known allergy to study medications
* Chronic opioid consumption (>3 months)
* Currently using lidocaine patches
* Pre-existing neuropathy
* A history of CVA
* High grade atrioventricular block (cardiac conduction system impairment)
* Organ dysfunction (cardiac failure, respiratory failure, end stage renal disease, hepatic dysfunction, hypoalbuminemia)
* Morbid obesity (≥40 kg/m2)
* Prior surgery in supra and/or infrainguinal region
* Non-English-speaking participants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time of administration of first analgesic after the surgery | Time to first analgesic request, defined as the interval (in minutes) from block administration to the first request for rescue analgesia, assessed for up to 24 hours.

SECONDARY OUTCOMES:
Total opioid consumption (converted to morphine milligram equivalents) | From the start of surgery through 48 hours postoperatively
  Intraoperative period; PACU; and at 6, 12, 24, and 48 hours following surgery.
Quality of Recovery | 24 hours
  The QoR-15 questionnaire has 15 questions that assess patient-reported quality of a patient's postoperative recovery using a 11-point numerical rating scale that leads to a minimum score of 0 (poor recovery) and a maximum score of 150 (excellent recovery).
Pain Scores | Up to two hours [post anesthesia recovery unit], 6 hours, 12 hours, 24 hours and 48 hours after surgery
  Patients will be asked to rate their pain score on a 11-point scale (0 = no pain to 10 = excruciating pain).

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez Martin MT, Alvarez Lopez S, Aldecoa Alvarez-Santullano C. Role of adjuvants in regional anesthesia: A systematic review. Rev Esp Anestesiol Reanim (Engl Ed). 2023 Feb;70(2):97-107. doi: 10.1016/j.redare.2021.06.006. Epub 2023 Feb 20. PMID 36813032
- [Background] Chen A, Duan W, Hao R, Wang C, Xu X. Ultrasound-guided dexmedetomidine combination with modified high fascia iliaca compartment block for arthroscopic knee surgery: what is the optimal dose of dexmedetomidine? BMC Anesthesiol. 2023 Dec 6;23(1):400. doi: 10.1186/s12871-023-02361-0. Erratum In: BMC Anesthesiol. 2023 Dec 22;23(1):421. doi: 10.1186/s12871-023-02391-8. PMID 38057762
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800